CLINICAL TRIAL: NCT04569474
Title: Efficacy of Sterile Dressing in the Prevention of of Peripheral Intravenous Catheters Associated Phlebitis in Patients From the Western Brazilian Amazon: Pragmatic, Randomized, Blinded and Controlled Trail
Brief Title: Peripheral IV Dressing and Phlebitis in Patients From Amazon
Acronym: IVDRESAMAZON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Mavilde da Luz Gonçalves Pedreira, Professor; supervisor of Sandra Maria Sampaio Enes, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2198630
Record Dates: First submitted 2018-04-02; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Phlebitis; Catheter Complications
MeSH Terms: conditions — Phlebitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dressing Group (Experimental): use of sterile transparent dressing
  Interventions: Device: Transparent dressing
- Standard Group (No Intervention): non-sterile transparente dressing

INTERVENTIONS:
Device: Transparent dressing — Use of sterile transparente dressing
  Arms: Dressing Group

SUMMARY:
Pragmatic, randomized, single-blinded, controlled clinical trial of the effect of dressing and stabilization of peripheral intravenous catheters on the occurrence of phlebitis in adult patients attended at a hospital from the Western Brazilian Amazon.

DETAILED DESCRIPTION:
Peripheral venous catheterization is the most commonly performed invasive procedure in healthcare. Care practices and the use of technologies may influence the results of the use peripheral intravenous catheters (PIC), contributing to the reduction of complications and adverse events. Phlebitis is characterized as one of the most serious complication related to the use of PIC and this study has as hypothesis to analyze if the occurrence of phlebitis associated with PIC is influenced by the use of sterile dressing. Objectives: To verify the effect of using sterile dressing and sterile adhesive tape compared to non-sterile adhesive tape in PIC on the occurrence of phlebitis in adult patients attended at a hospital from the Western Brazilian Amazon. Methods: Pragmatic, randomized, controlled and single-blinded clinical study conducted in Rio Branco, Acre. The sample was calculated in 330 patients, aged 18 years or older and who met the inclusion criteria. Data collection took place between June 2018 and September 2019, after approval of ethical merit. To identify the type of sterile transparent dressing to be studied, was carried out an implementation study with a final sample of 71 patients, focusing analysis from the perspective of the patient, professional and clinics. The patients of the clinical study were randomly allocated to one of the study groups: Experimental group (sterile transparent dressing) or Standard Group (non-sterile adhesive tape). Phlebitis was diagnosed by the bedside nurse, according to presence and severity. If present, the nurse removed the CIP and an external evaluator was called to perform a diagnose of phlebitis with blindness regarding the intervention. Variables related to patient characterization, intravenous therapy, peripheral venipuncture, reasons for withdrawal and length of PIC stay, reasons for removal and length of coverage, and associated complications were investigated. For the statistical analysis, Chi-square, Fisher's Exact, student t test, and Mann-Whitney U tests were used. The multiple analysis was performed using the logistic regression model to estimate the Relative Risk (RR) and the Kaplan-Meier model, Cox regression, for survival analysis. RR calculation for 95% Confidence Interval (IC) was applied to estimate the degree of association between variables. In all tests, the significance level of 5% was considered.

ELIGIBILITY:
Inclusion Criteria:

* IV access for more 48 hours obtained in the studied wards.
* IV access 20 and 22 G.
* without confusion or agitation
* Aged more or equal 18 years

Exclusion Criteria:

* Sepsis
* Skin lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2018-05-06 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Phlebitis | Unitl day 7 of catheter placement and study participation
  Vein inflamation measure by Scale Grades from Infusion Nursing Society rating from zero (absence) to 4 (severe phlebitis)

CONTACTS AND LOCATIONS:
Overall Officials: Mavilde LG Pedreira, PhD, Principal Investigator — Full Professor
Locations (2):
- Brazil (2):
  - Federal University of São Paulo, São Paulo
  - Universidade Federal de São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-07-06): https://cdn.clinicaltrials.gov/large-docs/74/NCT04569474/Prot_000.pdf